CLINICAL TRIAL: NCT02749851
Title: Functional Imaging of Human Placenta by MRI
Brief Title: Placenta Imaging Project
Acronym: PIP
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Antonio E. Frias, Associate Professor, Oregon Health and Science University
Other Study IDs: OHSU IRB 15196; U01HD087182 (NIH)
Record Dates: First submitted 2016-02-08; First posted 2016-04-25 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: High Risk Pregnancy
Keywords: pregnancy; growth restriction
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens to be included:
  Maternal blood (10ml) taken at each MRI visit and prior to delivery Maternal urine taken at each MRI visit and prior to delivery Placental tissue collected at the time of delivery.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Non-smokers: Pregnant women that identify as non-smokers with low risk for placental insufficiency will receive the MRI Imaging intervention.
  Interventions: Device: MRI
- Smokers: Pregnant women that identify as smokers will receive the MRI Imaging intervention.
  Interventions: Device: MRI
- High risk/Non-Smokers: Pregnant women that identify as non-smokers who are at a high risk for adverse outcomes based on prior clinical history will receive the MRI Imaging intervention.
  Interventions: Device: MRI
- Confirmed IUGR: Pregnant women identified by their clinical care provided to have confirmed IUGR during their current pregnancy
  Interventions: Device: MRI - IUGR

INTERVENTIONS:
Device: MRI — Recently-developed placenta-specific magnetic resonance imaging (MRI) tools will be used to quantify maternal perfusion and oxygen transfer throughout pregnancy in 3 groups of human subjects: 1) non-smokers, 2) smokers, 3) individuals at high risk for adverse outcome. The objective of this work is to develop a new non-invasive clinical tool for early identification of placental dysfunction.
  Other Names: magnetic resonance imaging
  Groups: High risk/Non-Smokers; Non-smokers; Smokers
Device: MRI - IUGR — Recently-developed placenta-specific magnetic resonance imaging (MRI) tools will be used to quantify maternal perfusion and oxygen transfer throughout pregnancy. The objective of this ancillary arm is to further test the sensitivity of placental magnetic resonance imaging to detect abnormal perfusion and oxygenation in confirmed cases of IUGR between gestational ages 28 to 36 weeks.
  Other Names: magnetic resonance imaging
  Groups: Confirmed IUGR

SUMMARY:
The purpose of this study is to test the application of newly generated magnetic resonance imaging (MRI) protocols for the assessment of placental perfusion in human subjects. The primary objective is to validate and establish the utility of placental MRI in pregnant women. The study will be entirely MRI-technology based with collection of placental tissue at the time of infant delivery for later correlative studies.

DETAILED DESCRIPTION:
The placenta provides all the nutrition from a pregnant mother to a developing fetus. A placenta that functions normally is needed to ensure normal fetal growth and development. Unfortunately, the placenta is the least understood human organ even though it is involved in all pregnancy complications. The placenta is so poorly understood because our current methods to look at it during pregnancy, like ultrasound, do not provide enough information about placental growth and function.

This study will help provide information about:

* How the placenta grows and develops during pregnancy
* How the placenta delivers nutrients, like oxygen to the developing fetus
* If placental function using new advanced imaging tools can predict pregnancy complications like fetal growth restriction, stillbirth, preeclampsia and preterm labor

This study will explore how blood flow to the placenta affects placental growth, fetal growth, and oxygen delivery to the fetus. Blood flow to the placenta may determine how the placenta supports fetal growth and development. Having a way to measure placental function during pregnancy may provide a way to understand normal pregnancies but importantly also identify pregnancies at increased risk for pregnancy complications.

Additionally we want to have an ancillary intrauterine growth restriction (IUGR) arm; the objective of this ancillary study is to test the sensitivity of the placental MRI protocol in women with confirmed cases of IUGR in the third trimester.

ELIGIBILITY:
Pregnant women will be recruited based on inclusion criteria for 3 subject groups:

1. Non-smokers with low risk for placental insufficiency
2. Smokers
3. Non-smokers who are at a high risk for adverse outcomes based on prior clinical history.

Inclusion criteria: Pregnant women fulfilling inclusion criteria, and not meeting exclusion criteria, will be invited to participate in this study.

Inclusion criteria for all groups:

1. Maternal age over 18 years and able to give informed consent
2. Pregnant patient, as defined by positive pregnancy test for elevated β-human chorionic gonadotropin (HCG) and certain menstrual history, or early ultrasound, identified prior to 14 weeks of gestation

Inclusion criteria for low risk group:

1. No history of a second or third trimester loss
2. No history of fetal growth restriction

Inclusion criteria for high risk group:

1. History of pregnancy complicated by placental insufficiency in a previous singleton pregnancy (i.e. severe preeclampsia requiring preterm delivery, preterm delivery due to placenta insufficiency (eg. fetal growth restriction (FGR), oligohydramnios, abnormal umbilical artery Doppler's, abnormal antenatal testing), FGR <10% delivered at term; stillbirth attributed to placental cause, regardless of gestational age
2. Not currently a smoker
3. Pregnancy at risk for placental insufficiency due to clinical concerns (eg. chronic hypertension)
4. Spontaneous preterm birth <34 weeks

Exclusion criteria: These criteria will exclude women whose medications, personality traits or obstetric conditions could confound their ability to complete a 1 hour MRI scan.

1. Individuals with intellectual disability or who are incarcerated
2. Multiple gestation
3. Major fetal anomalies known to be associated with abnormal growth (i.e. major congenital heart defect, gastroschisis)
4. Current maternal history of alcohol or illicit drug use
5. Current medical problems requiring chronic treatment:

   * Cancer
   * Active liver disease (acute hepatitis, chronic active hepatitis, persistently abnormal liver enzymes)
   * Chronic pulmonary disease including asthma requiring regular use of medication
6. Prior history of claustrophobia
7. Metal implants
8. Increased aneuploidy risk based on ultrasound findings or genetic testing

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who plan to deliver at OHSU or University of Utah hospitals and live within the areas served by those medical facilities.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Placental perfusion (Units of measure: ml/min) measured at 3 time points across gestation. | Change from 16, 24, and 32 weeks gestation
  This will allow perfusion changes across pregnancy to be quantified in women from the three study groups.
Optimal cutoff values of placental MRI for placenta mediated adverse outcomes using receiver operating characteristics (ROC) | Change from 16, 24, and 32 weeks gestation
  Determine the sensitivity and specificity of placental MRI at 16, 24, and 32 weeks gestation for identifying risk of adverse clinical outcome identified later in pregnancy. Optimal cutoff values of placental MRI for placenta mediated adverse outcomes using receiver operating characteristics (ROC).
Composite of placenta-mediated adverse pregnancy outcomes | 39 weeks gestation
  A binary variable indication whether the placenta-mediated adverse pregnancy has observed within 39 weeks gestation
  Composite of placenta-mediated adverse pregnancy outcomes defined as the presence of at least one of the following:
  1. Fetal death (not due to genetic or infectious etiology),
  2. Preeclampsia or gestational hypertension,
  3. Small for gestational age fetus < 5%,
  4. Oligohydramnios (defined as amniotic fluid index (AFI) < 5 cm) prompting delivery prior to 39 weeks gestation,
  5. Abnormal fetal heart rate tracing prompting delivery prior to 39 weeks gestation,
  6. Abnormal umbilical artery Doppler velocimetry prompting delivery prior to 39 weeks gestation.

SECONDARY OUTCOMES:
Composite of Placenta histologic outcomes | 39 weeks gestation
  Composite of placental histologic outcomes defined as the presence of one of the following:
  1. accelerated villous maturation
  2. abnormal villous cytotrophoblast proliferation
  3. microscopic infarctions
  4. decidual vasculopathy
Diagnosis of preeclampsia using standard clinical criteria | 39 weeks gestation
Small for gestational age fetus at 3% and 5% | 39 weeks gestation
Gestational age at delivery prior to 37 weeks gestation. | 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Frias, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schabel MC, Roberts VHJ, Gibbins KJ, Rincon M, Gaffney JE, Streblow AD, Wright AM, Lo JO, Park B, Kroenke CD, Szczotka K, Blue NR, Page JM, Harvey K, Varner MW, Silver RM, Frias AE. Quantitative longitudinal T2* mapping for assessing placental function and association with adverse pregnancy outcomes across gestation. PLoS One. 2022 Jul 19;17(7):e0270360. doi: 10.1371/journal.pone.0270360. eCollection 2022. PMID 35853003